CLINICAL TRIAL: NCT02280928
Title: Development and Evaluation of a Home-Based Dual-Task Training Program to Improve Balance Performance for Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chiang Mai University (Other)
Responsible Party: Principal Investigator, Patima Silsupadol, Faculty of Associated Medical Sciences, Chiang Mai University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: The graduate school, CMU
Record Dates: First submitted 2014-10-30; First posted 2014-11-03 (Estimated); Last update posted 2015-07-22 (Estimated); Status verified 2015-07

CONDITIONS: Elderly; Aged
MeSH Terms: interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Single-task motor training group (Experimental): The participants will receive only balance training which will progress from stance activities, to stance activities plus hand manipulation, then gait activities, and finally gait activities plus hand manipulation.
  Interventions: Other: Balance exercise
- Single-task cognitive training group (Experimental): The participants will receive cognitive training that will involve executive function, attention, and working memory.
  Interventions: Other: Cognitive training
- Dual-task motor-cognitive training group (Experimental): The participants assigned to the dual-task motor-cognitive training group will receive the same exercises as single-task motor training while simultaneously performing secondary tasks as those in the single-task cognitive training group.
  Interventions: Other: Balance exercise; Other: Cognitive training
- Dual-task cognitive-cognitive training group (Experimental): The participants in the dual-task cognitive-cognitive trainings group will receive two cognitive tasks at the same time.
  Interventions: Other: Dual-task cognitive-cognitive training

INTERVENTIONS:
Other: Balance exercise — Balance activities, using a task-oriented approach, progress participants from body stability, to body stability plus hand manipulation, then body transport, and finally body transport plus hand manipulation.
  Arms: Dual-task motor-cognitive training group; Single-task motor training group
Other: Cognitive training — Cognitive training involves executive function, attention, and working memory. Examples of cognitive training include finding the exit to a maze, calculation, visual-spatial skills, Sudoku, Stroop color-word task, word search, spot the differences, visual discrimination, and memory scanning skills.
  Arms: Dual-task motor-cognitive training group; Single-task cognitive training group
Other: Dual-task cognitive-cognitive training — The Dual-task cognitive-cognitive training involves applying two cognitive tasks at the same time.
  Arms: Dual-task cognitive-cognitive training group

SUMMARY:
The purpose of this study is to (1) develop and test the effectiveness of home-based interventions on dual-task performance in older adults; and (2) determine the generalizability of the four trainings (i.e. single-task motor training, single-task cognitive training, dual-task motor-cognitive training, and dual-task cognitive-cognitive trainings) to novel tasks.

DETAILED DESCRIPTION:
Although, dual-task motor-cognitive training has proven to be more effective in improving dual-task balance performance than traditional single-task motor training, poor evidence of training-related transfer to a novel dual task has been shown. Additionally, another important impediment to the development of intervention to improve dual-task balance performance is that the previous studies have largely focused on training in a laboratory, or clinical setting, often with one-on-one supervision by a therapist or research assistant. Even though the home-based approach is more pragmatic, desirable, and encourages accessibility, no study has been done to examine the efficacy of home-based dual-task training.

Therefore, this study aims to address these gaps in the literature by conducting a home-based program designed to improve dual-task performance with a broader transfer-of-training effects in older adults. Participants will be randomly assigned to one of four groups (i.e. single-task motor training, single-task cognitive training, dual-task motor-cognitive training, and dual-task cognitive-cognitive trainings).

ELIGIBILITY:
Inclusion Criteria:

* Able to walk at least 10 meters without any assistive device
* Having greater than 16/23 for illiterate persons, greater than 20/30 for primary education level persons, and greater than 23/30 for secondary education level persons on the Mini-Mental State Examination-Thai 2002 (MMSE-Thai2002)

Exclusion Criteria:

* Severe neurological problems that could account for possible imbalance such as cerebral vascular accident, Parkinson's disease, transient ischemic attacks, and neuropathy
* Severe musculoskeletal problems that could impact gait such as severe osteoarthritis and active inflammatory joint disease
* Severe cardiopulmonary problems such as asthma and chronic obstructive pulmonary disease
* Visual impairment that cannot be corrected by lenses
* Severe auditory impairment such as deafness
* Depression as scored ≥ 13 by Thai Geriatric Depression Scale (TGDS)

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
The Center of Mass velocity and Base of Support distance | At baseline and after 4-week training
  The Center of Mass velocity and Base of Support distance is referred as the direction of the center of mass velocity in relation to base of support. It is used to measure the control of dynamic balance throughout gait under single-task and dual-task conditions in order to examine training effect.
Spatio-temporal gait parameters | At baseline and after 4-week training
  Spatio-temporal gait parameters is measured throughout gait under single-task and dual-task conditions in order to examine training effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Associated Medical Sciences, Chiang Mai University, Sripoom, Chiang Mai, Thailand